CLINICAL TRIAL: NCT02909686
Title: Effects of Botanical Microglia Modulators in Gulf War Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jarred Younger, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: F150318011; CDMRP-GW130015 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Gulf War Illness
Keywords: Gulf War Syndrome; Chronic Multisymptom Illnesses; Medically Unexplained Illnesses
MeSH Terms: conditions — Persian Gulf Syndrome | interventions — Frankincense; Curcumin; turmeric extract; fisetin; Luteolin; stinging nettle lectin; pycnogenols; Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Boswellia Serrata (Experimental): 400-800mg in capsule form by mouth every day
  Interventions: Dietary Supplement: Boswellia Serrata
- Curcumin (Experimental): 1000-2000mg in capsule form by mouth every day
  Interventions: Dietary Supplement: Curcumin
- Epimedium (Experimental): 1000-2000mg in capsule form by mouth every day
  Interventions: Dietary Supplement: Epimedium
- Fisetin (Experimental): 200-800mg in capsule form by mouth every day
  Interventions: Dietary Supplement: Fisetin
- Luteolin (Experimental): 200-400mg in capsule form by mouth every day
  Interventions: Dietary Supplement: Luteolin
- Nettle (Experimental): 435-1305mg in capsule form by mouth every day
  Interventions: Dietary Supplement: Nettle
- Pycnogenol (Experimental): 200-400mg in capsule form by mouth every day
  Interventions: Dietary Supplement: Pycnogenol
- Reishi Mushroom (Experimental): 1600-3200mg in capsule form by mouth every day
  Interventions: Dietary Supplement: Reishi Mushroom
- Resveratrol (Experimental): 200-600mg in capsule form by mouth every day
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): in capsule form by mouth every day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Boswellia Serrata
  Other Names: Indian frankincense
  Arms: Boswellia Serrata
Dietary Supplement: Curcumin
  Other Names: Curcumasorb; Turmeric extract; Meriva
  Arms: Curcumin
Dietary Supplement: Epimedium
  Other Names: Barrenwort; Bishop's Hat; Fairy Wings; Horny Goat Weed; Yin Yang Huo
  Arms: Epimedium
Dietary Supplement: Fisetin
  Arms: Fisetin
Dietary Supplement: Luteolin
  Arms: Luteolin
Dietary Supplement: Nettle
  Other Names: Common Nettle; urtica dioica; Stinging Nettle
  Arms: Nettle
Dietary Supplement: Pycnogenol
  Other Names: Maritime Pine Extract; Pine Bark Extract
  Arms: Pycnogenol
Dietary Supplement: Reishi Mushroom
  Arms: Reishi Mushroom
Dietary Supplement: Resveratrol
  Other Names: Red Wine Extract
  Arms: Resveratrol
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The overall objective of this protocol is to test if Gulf War Illness (GWI) involves chronic inflammation that cannot be measured with typical techniques. The investigators will be observing the effects of nine different botanical compounds (supplements) that are known to suppress inflammation. If one of those supplements helps the symptoms of GWI, it will give the investigators information about what is wrong in people with GWI.

DETAILED DESCRIPTION:
There is still a poor understanding of the pain, fatigue, and other symptoms that affect approximately 250,000 veterans. The precise mechanism of Gulf War Illness (GWI) is not understood, and there is no targeted treatment for the condition. A current model for GWI points to the central nervous system, immune cells, called microglia that may be hyperactive in patients with GWI. Discovering effective treatments for this disorder is a top priority of GWI research.

Given the investigator's preliminary data, it is suspected that GWI is a form of low-level neuroinflammation that involves hypersensitivity of receptors on microglia. In order to help test that hypothesis, the investigators will be administering supplements that have been shown in vitro or animal in vivo to suppress microglia function in a way that is anti-inflammatory and neuroprotective. If any of these agents suppress symptoms in GWI, it will give the investigators important information about the disease that may allow for creation of better diagnostic tools and treatments in future research studies. Observing the effects of the selected nine anti-inflammatory botanical compounds, in this clinical study, is a strong compliment to the ongoing mechanistic GWI research.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age 39-65, inclusive
3. Veterans who meet the Kansas inclusion criteria for GWI
4. Present in Persian Gulf between 1990 and August 1991
5. Patient completes daily report during 2 week baseline period (at least 80% completion rate)
6. Able to receive a venous blood draw

Exclusion Criteria:

1. Positive rheumatoid factor at screening
2. Positive anti-nuclear antibody at screening
3. C-reactive protein> 3mg/L at screening
4. Erythrocyte Sedimentation Rate> 40mm/hr at screening
5. Auto-immune disorder
6. Diagnosed Rheumatologic Condition
7. Major PTSD symptoms
8. Hypotension (under 90/60 mm Hg) or history of cardiovascular disease
9. Antihypertensive, anticoagulant medication, nitroglycerine, lithium medication use
10. Diabetes with Hemoglobin A1C >9%
11. History of anaphylaxis to study botanical compounds
12. Current daily use of opioid medication
13. Hospital Anxiety and Depression Scale, Depression subscale score of 16 or higher at baseline
14. Current litigation of worker's compensation claim
15. Blood or clotting disorder
16. Acute infection (body temperature over 100 degrees F)
17. Current daily use of confounding-anti-inflammatory medication as part of regular medication regimen
18. Individuals that are not able to read & understand English

Ages: 39 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2022-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jarred W Younger, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Younger J, Donovan EK, Hodgin KS, Ness TJ. A Placebo-Controlled, Pseudo-Randomized, Crossover Trial of Botanical Agents for Gulf War Illness: Reishi Mushroom (Ganoderma lucidum), Stinging Nettle (Urtica dioica), and Epimedium (Epimedium sagittatum). Int J Environ Res Public Health. 2021 Apr 1;18(7):3671. doi: 10.3390/ijerph18073671. PMID 33915962
- [Derived] Hodgin KS, Donovan EK, Kekes-Szabo S, Lin JC, Feick J, Massey RL, Ness TJ, Younger JW. A Placebo-Controlled, Pseudo-Randomized, Crossover Trial of Botanical Agents for Gulf War Illness: Resveratrol (Polygonum cuspidatum), Luteolin, and Fisetin (Rhus succedanea). Int J Environ Res Public Health. 2021 Mar 3;18(5):2483. doi: 10.3390/ijerph18052483. PMID 33802381
- [Derived] Donovan EK, Kekes-Szabo S, Lin JC, Massey RL, Cobb JD, Hodgin KS, Ness TJ, Hangee-Bauer C, Younger JW. A Placebo-Controlled, Pseudo-Randomized, Crossover Trial of Botanical Agents for Gulf War Illness: Curcumin (Curcuma longa), Boswellia (Boswellia serrata), and French Maritime Pine Bark (Pinus pinaster). Int J Environ Res Public Health. 2021 Mar 3;18(5):2468. doi: 10.3390/ijerph18052468. PMID 33802272

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants took as least one botanical. Some then went on to take a second or even third botanical, but not all participants did this. The order was randomized, so not all participants took the same sequence of botanicals.
Pre-assignment Details: Participants also took a placebo for each botanical. The order is as follows for each botanical: 30 +/- 3 days pf baseline symptom reports, followed by 30+/- days of placebo, followed by 30+/- days days of lower-dose botanical, followed by 30+/- days of higher-dose botanical.
Groups:
- All Participants: Participants enrolled in this study were assigned to receive placebo and up to three botanical agents in a psuedo-randomized order. For each botanical condition, participants first received a placebo, followed by a lower dose of botanical and a higher dose of botanical, for up to three different botanicals. After completing the full protocol of three botanicals, participants were then offered the opportunity to re-enroll to receive up to three additional botanicals.
  Dietary Supplement: Boswellia Serrata 400-800mg in capsule form by mouth every day Dietary Supplement: Curcumin 1000-2000mg in capsule form by mouth every day Dietary Supplement: Epimedium 1000-2000mg in capsule form by mouth every day Dietary Supplement: Fisetin 200-800mg in capsule form by mouth every day Dietary Supplement: Luteolin 200-400mg in capsule form by mouth every day Dietary Supplement: Nettle 435-1305mg in capsule form by mouth every day Dietary Supplement: Pycnogenol 200-400mg in capsule form by mouth every day Dietary Supplement: Reishi 1600-3200mg in capsule form by mouth every day Dietary Supplement: Resveratrol 200-600mg in capsule form by mouth every day Dietary Supplement: Placebo in capsule form by mouth every day
Period: Overall Study
Arm/Group | All Participants
Started | 96
Boswellia Serrata | 10
Curcumin | 10
Epimedium | 11
Fisetin | 11
Luteolin | 11
Nettle | 12
Pycnogenol | 11
Reishi Mushroom | 10
Resveratrol | 10
Placebo | 96
Completed | 91
Not Completed | 5
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Participants enrolled in this study were assigned to receive placebo and up to three botanical agents in a psuedo-randomized order. For each botanical condition, participants first received a placebo, followed by a lower dose of botanical and a higher dose of botanical, for up to three different botanicals. After completing the full protocol of three botanicals, participants were then offered the opportunity to re-enroll to receive up to three additional botanicals.
Groups:
- All Participants: Participants enrolled in this study were assigned to receive placebo and up to three botanical agents in a psuedo-randomized order. For each botanical condition, participants first received a placebo, followed by a lower dose of botanical and a higher dose of botanical, for up to three different botanicals. After completing the full protocol of three botanicals, participants were then offered the opportunity to re-enroll to receive up to three additional botanicals
Arm/Group | All Participants
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Overall Gulf War Illness Disease Severity
Description: Self reported Gulf War Illness symptom severity evening reports were collected for the duration of the study. Scale= change from baseline in overall GWI Disease severity (-100 to +100, with positive numbers indicating how much the symptom improved).
Time Frame: Week 17
Population: Participants assigned to multiple arms
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Boswellia Serrata: 400-800mg in capsule form by mouth every day
  Boswellia Serrata
- Curcumin: 1000-2000mg in capsule form by mouth every day
  Curcumin
- Epimedium: 1000-2000mg in capsule form by mouth every day
  Epimedium
- Fisetin: 200-800mg in capsule form by mouth every day
  Fisetin
- Luteolin: 200-400mg in capsule form by mouth every day
  Luteolin
- Nettle: 435-1305mg in capsule form by mouth every day
  Nettle
- Pycnogenol: 200-400mg in capsule form by mouth every day
  Pycnogenol
- Reishi Mushroom: 1600-3200mg in capsule form by mouth every day
  Reishi Mushroom
- Resveratrol: 200-600mg in capsule form by mouth every day
  Resveratrol
- Placebo: in capsule form by mouth every day
  Placebo
Arm/Group | Boswellia Serrata | Curcumin | Epimedium | Fisetin | Luteolin | Nettle | Pycnogenol | Reishi Mushroom | Resveratrol | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 9 | 89
units on a scale | 13 (.43) | 0 (.32) | 8 (1.56) | -1 (2.08) | 12 (.90) | 19 (1.08) | 15 (1.18) | -5 (2.08) | 14 (1.1) | 7 (1.37)

2. Secondary Outcome: Change From Baseline in Pain Severity
Description: Self reported pain symptom severity evening reports were collected for the duration of the study. Scale= change from baseline in overall GWI pain severity (-100 to +100, with positive numbers indicating how much the symptom improved).
Time Frame: Week 17
Population: Participants assigned to multiple arms
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Boswellia Serrata | Curcumin | Epimedium | Fisetin | Luteolin | Nettle | Pycnogenol | Reishi Mushroom | Resveratrol | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 9 | 89
units on a scale | 13 (1.12) | -1 (.95) | 8 (1.15) | 1 (1.87) | 11 (.94) | 14 (1.35) | 13 (1.07) | -2 (1.53) | 13 (1.42) | 6 (1.31)

3. Secondary Outcome: Change From Baseline in Fatigue Severity
Description: Self reported fatigue symptom severity evening reports were collected for the duration of the study. Scale= change from baseline in overall GWI fatigue severity (-100 to +100, with positive numbers indicating how much the symptom improved).
Time Frame: Week 17
Population: Participants assigned to multiple arms
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Boswellia Serrata | Curcumin | Epimedium | Fisetin | Luteolin | Nettle | Pycnogenol | Reishi Mushroom | Resveratrol | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 9 | 89
units on a scale | 6 (2.01) | 4 (1.89) | 4 (1.89) | -5 (1.99) | 11 (1.81) | 4 (2.60) | 3 (2.03) | 3 (0.67) | 10 (1.62) | 4 (1.46)

4. Secondary Outcome: Change From Baseline in Cognitive Symptom Severity
Description: Self reported Cognitive Symptom Severity evening reports were collected for the duration of the study. Scale= change from baseline in overall Cognitive Symptom Severity (-100 to +100, with positive numbers indicating how much the symptom improved).
Time Frame: Week 17
Population: Participants assigned to multiple arms
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Boswellia Serrata | Curcumin | Epimedium | Fisetin | Luteolin | Nettle | Pycnogenol | Reishi Mushroom | Resveratrol | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 9 | 89
units on a scale | -6 (2.2) | 7 (0.70) | 0 (1.94) | 3 (2.25) | -4 (1.76) | -11 (1.34) | -8 (1.71) | -1 (2.33) | -9 (1.61) | -4 (1.57)

5. Secondary Outcome: Change From Baseline in Mood Symptom Severity
Description: Self reported Mood Symptom Severity evening reports were collected for the duration of the study. Scale= change from baseline in overall Mood Symptom Severity (-100 to +100, with positive numbers indicating how much the symptom improved).
Time Frame: Week 17
Population: Participants assigned to multiple arms
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Boswellia Serrata | Curcumin | Epimedium | Fisetin | Luteolin | Nettle | Pycnogenol | Reishi Mushroom | Resveratrol | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 9 | 89
units on a scale | 7 (1.84) | 12 (1.1) | 6 (1.94) | 0 (1.42) | 1 (1.74) | -9 (0.99) | -7 (1.26) | 0 (0.02) | -3 (1.63) | 1 (1.53)

6. Secondary Outcome: Change From Baseline in Dermatological Symptom Severity
Description: Self reported Dermatological Symptom Severity evening reports were collected for the duration of the study. Scale= change from baseline in overall Dermatological Symptom Severity (-100 to +100, with positive numbers indicating how much the symptom improved).
Time Frame: Week 17
Population: Participants assigned to multiple arms
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Boswellia Serrata | Curcumin | Epimedium | Fisetin | Luteolin | Nettle | Pycnogenol | Reishi Mushroom | Resveratrol | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 9 | 89
units on a scale | 3 (0.38) | -4 (0.29) | -3 (0.29) | 0 (0.75) | 1 (0.55) | 1 (0.48) | 3 (0.42) | -2 (1.14) | 2 (0.51) | 0 (0.57)

7. Secondary Outcome: Change From Baseline in Respiratory Symptom Severity
Description: Self reported Respiratory Symptom Severity evening reports were collected for the duration of the study. Scale= change from baseline in overall Respiratory Symptom Severity (-100 to +100, with positive numbers indicating how much the symptom improved).
Time Frame: Week 17
Population: Participants assigned to multiple arms
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Boswellia Serrata | Curcumin | Epimedium | Fisetin | Luteolin | Nettle | Pycnogenol | Reishi Mushroom | Resveratrol | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 9 | 89
units on a scale | -3 (0.91) | -1 (1.07) | -5 (0.42) | 0 (1.15) | 3 (0.59) | -2 (0.50) | -1 (0.66) | 0 (1.08) | 1 (0.67) | 0 (0.66)

8. Secondary Outcome: Change From Baseline in Gastrointestinal Symptom Severity
Description: Self reported Gastrointestinal Symptom Severity evening reports were collected for the duration of the study. Scale= change from baseline in overall Gastrointestinal Symptom Severity (-100 to +100, with positive numbers indicating how much the symptom improved).
Time Frame: Week 17
Population: Participants assigned to multiple arms
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Boswellia Serrata | Curcumin | Epimedium | Fisetin | Luteolin | Nettle | Pycnogenol | Reishi Mushroom | Resveratrol | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 9 | 89
units on a scale | 9 (0.39) | -5 (2.04) | -2 (1.37) | 8 (0.85) | 6 (0.66) | 1 (1.07) | 4 (0.84) | -12 (1.20) | 1 (1.48) | 1 (1.18)

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Boswellia Serrata | Curcumin | Epimedium | Fisetin | Luteolin | Nettle | Pycnogenol | Reishi Mushroom | Resveratrol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/11 | 0/11 | 0/12 | 0/11 | 0/10 | 0/10 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/11 | 0/11 | 0/12 | 0/11 | 0/10 | 0/10 | 0/96
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/11 | 0/11 | 1/12 | 0/11 | 0/10 | 0/10 | 0/96
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boswellia Serrata (N=10) | Curcumin (N=10) | Epimedium (N=11) | Fisetin (N=11) | Luteolin (N=11) | Nettle (N=12) | Pycnogenol (N=11) | Reishi Mushroom (N=10) | Resveratrol (N=10) | Placebo (N=96)
Elevated Liver Enzyme (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT02909686/Prot_SAP_000.pdf